CLINICAL TRIAL: NCT03110575
Title: A 12-Week Open-Label Extension Study to Evaluate TNX-102 SL Taken Daily at Bedtime in Patients With PTSD
Brief Title: 12-Week Open-Label Extension Study of TNX-102 SL in PTSD Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped early due to inadequate separation on primary efficacy endpoint in the lead-in HONOR study, TNX-CY-P301
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-P303
Record Dates: First submitted 2017-03-31; First posted 2017-04-12 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: PTSD
Keywords: TNX-102 SL; Bedtime; Sublingual; 3-month; Safety; Efficacy; PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TNX-102 SL (Experimental): 2 x TNX-102 SL, 2.8 mg tablets taken daily at bedtime for 12 weeks
  Interventions: Drug: TNX-102 SL

INTERVENTIONS:
Drug: TNX-102 SL — 2 x TNX-102 SL, 2.8mg tablets taken daily at bedtime for 12 weeks
  Other Names: cyclobenzaprine HCl

SUMMARY:
This is an open-label, extension trial designed to evaluate safety over 12 additional weeks of TNX-102 SL therapy taken daily at bedtime for the treatment of PTSD. Patients recruited into this trial are those who have successfully completed the double-blind lead-in study.

DETAILED DESCRIPTION:
The study will consist of 5 study visits, including Screening/Baseline Visit 1 (Day 0, which is anticipated to be the same visit as the last visit on double-blind treatment), a phone visit after 2 weeks of treatment, and in-clinic visits after 4, 8, and 12 weeks of treatment.

The primary objective of the study is to evaluate the safety of TNX-102 SL tablets taken daily at bedtime over an additional 12 weeks in patients with PTSD who have completed a double-blinded lead-in study.

The secondary objective of the study is to evaluate the efficacy of TNX-102 SL tablets taken daily at bedtime over an additional 12 weeks in patients with PTSD who have completed a double-blinded lead-in study.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed the final treatment study visit of the lead-in study and remained compliant with the lead-in protocol and study treatment.
* The patient has provided written informed consent to participate in this extension protocol.
* Female patients of childbearing potential continue to agree to practice one of the medically acceptable methods of birth control detailed in the lead-in study.

Exclusion Criteria:

* None.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Bedoya, Study Director — Premier Research
Locations (31):
- United States (31):
  - Phoenix, Phoenix, Arizona
  - Rogers, Rogers, Arkansas
  - Beverly Hills, Beverly Hills, California
  - Glendale, Glendale, California
  - Oakland, Oakland, California
  - Oceanside, Oceanside, California
  - Orange, Orange, California
  - Riverside, Riverside, California
  - San Diego, San Diego, California
  - Temecula, Temecula, California
  - Colorado Springs, Colorado Springs, Colorado
  - Jacksonville, Jacksonville, Florida
  - Lake City, Lake City, Florida
  - Lauderhill, Lauderhill, Florida
  - Tampa, Tampa, Florida
  - Atlanta, Atlanta, Georgia
  - New Bedford, New Bedford, Massachusetts
  - Flowood, Flowood, Mississippi
  - Las Vegas, Las Vegas, Nevada
  - Berlin, Berlin, New Jersey
  - Cedarhurst, Cedarhurst, New York
  - New York, New York, New York
  - Canton, Canton, Ohio
  - Cincinnati, Cincinnati, Ohio
  - Dayton, Dayton, Ohio
  - Oklahoma City, Oklahoma City, Oklahoma
  - Charleston, Charleston, South Carolina
  - Austin, Austin, Texas
  - Dallas, Dallas, Texas
  - Houston, Houston, Texas
  - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo - TNX-102 SL: The patients in this group received placebo in the lead-in double blind study TNX-CY-P301, then received TNX-102 SL 5.6 mg in this open label study TNX-CY-P303.
- TNX-102 SL - TNX-102 SL: The patients in this group received TNX-102 SL 5.6 mg in the lead-in double blind study TNX-CY-P301, then received TNX-102 SL 5.6 mg in this open label study TNX-CY-P303.
Period: Overall Study
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
Started | 97 | 93
Completed | 68 | 67
Not Completed | 29 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL | Total
Number analyzed (Participants) | 97 | 93 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.19) | 36.1 (7.85) | 36.3 (8.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 82 | 87 | 169
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 34
  Not Hispanic or Latino | 79 | 77 | 156
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 4 | 6
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 17 | 22 | 39
  White | 64 | 56 | 120
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 97 | 93 | 190

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Newly Emergent Adverse Events of TNX-102 SL Tablets Taken Daily at Bedtime Over an Additional 12 Weeks in Patients With PTSD Who Have Completed a Double-blinded lead-in Study
Description: Adverse events will be coded using the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized overall and by preferred term and system organ class.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
Number analyzed (Participants) | 97 | 93
Participants | 62 | 40

2. Secondary Outcome: Change From Both Baselines in the Total Clinician Administered PTSD Scale for DSM-5 (CAPS-5) Score
Description: The CAPS-5 symptom severity 1-week recall version will be administered by qualified and trained clinicians. Score ranges from 0 to 80 with lower scores indicating less severe PTSD symptoms.
Time Frame: Day 1 of TNX-CY-P301 (Week -12 of TNX-CY-P303), Day 1 of TNX-CY-P303, Week 12 of TNX-CY-P303
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
Number analyzed (Participants) | 97 | 93
units on a scale
  Change from TNX-CY-P301 baseline | -24.5 (2.43) | -24.2 (2.64)
  Change from TNX-CY-P303 baseline | -6.2 (1.63) | -6.2 (1.78)

ADVERSE EVENTS:
Time Frame: 12 Weeks
Arm/Group | Placebo - TNX-102 SL | TNX-102 SL - TNX-102 SL
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/93
Other Adverse Events (participants affected / at risk) | 49/97 | 19/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo - TNX-102 SL (N=97) | TNX-102 SL - TNX-102 SL (N=93)
Hypoaesthesia Oral (Gastrointestinal disorders) | 29 | 12
Glossodynia (Gastrointestinal disorders) | 9 | 2
Paraesthesia oral (Gastrointestinal disorders) | 7 | 2
Somnolence (Nervous system disorders) | 9 | 8
Product Taste Abnormal (Product Issues) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT03110575/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03110575/SAP_001.pdf